CLINICAL TRIAL: NCT04343131
Title: The Effect of Three Different Types of Diet on Glycemia Assessed by Continuous Glucose Monitoring in Patients With Type 1 Diabetes on Multiple Daily Insulin Treatment
Brief Title: Different Dietary Interventions and Glycemia in T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Diet in T1DM
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Glycemia; Continuous glucose monitoring; Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean diet (Active Comparator): Mediterranean diet for 7 days
  Interventions: Behavioral: Dietary intervention
- Low-carb/high protein diet (Active Comparator): Low-carb/high protein diet for 7 days
  Interventions: Behavioral: Dietary intervention
- Reference diet (Active Comparator): Reference diet for 7 days
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Behavioral: Dietary intervention — Crossover dietary manipulation using three different types of diet for 7 days each

SUMMARY:
The aim of the present study was to compare the effects of three different dietary patterns on glycemia in individuals with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
The aim of the present crossover study was to compare the effects of three different dietary patterns on glycemia in individuals with type 1 diabetes (T1D).

Three different isocaloric diets, namely, a Mediterranean style diet, a low-carbohydrate diet and a reference diet were provided to patients with T1D for three separate weeks, in a random order, and with 7-day washout periods in-between. Glycemia was assessed during each 7-day period using a continuous glucose monitoring system. Participants were recruited from the outpatient diabetes clinic of a University Hospital in Athens, Greece.

The primary outcome was time spent in euglycaemic range (TIR: 70-140mg/dl) during the diet period. Secondary outcomes were: (a) time spent below euglycaemic range (TBR: <70mg/dl); (b) time spent above euglycaemic range (TAR: >140mg/dl); (c) glycaemic variability and (d) insulin needs.

ELIGIBILITY:
Inclusion Criteria:

* Adults with T1D receiving MDI therapy
* Sufficient education and knowledge on carbohydrate counting
* Motivation to follow a specific dietary schedule
* Frequent (7 times a-day) self-monitoring of blood glucose (SMBG)
* Willingness to wear a CGM system

Exclusion Criteria:

* HbA1c >8%
* Lack of severe diabetic complications, such as cardiovascular disease, proliferative retinopathy, nephropathy with estimated glomerular filtration rate (eGFR) ≤ 60 or gastroparesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent with glucose levels between 70-140 mg/dl | 7 days
  Percentage of time spent with glucose levels between 70-140 mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, MD, PhD, Principal Investigator — Medical School, National and Kapodistrian University of Athens, Laiko Hospital

IPD SHARING:
Plan to Share IPD: No